CLINICAL TRIAL: NCT01210287
Title: Incidence of HBV Reactivation in HBsAg Negative/HBcAb Positive Diffuse Large B Cell Lymphoma or High Grade Follicular Lymphoma Patients: A Prospective Study
Brief Title: Incidence of Hepatitis B Virus (HBV) Reactivation in HBsAg Negative/HBcAb Positive Lymphoma Patients Treated With RCHOP
Acronym: IHBVRL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junning Cao, Vice Director of the department of Medical Oncology, Fudan University Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 201010HBV
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Lymphoma
Keywords: hepatitis B virus reactivation; HBsAg negative; HBcAb positive; lymphoma; rituximab
MeSH Terms: conditions — Lymphoma | interventions — Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Observation (No Intervention): Observation of the HBV reactivation in HBsAg negative/HBcAg positive patients receiving RCHOP without prophylactic anti-HBV treatment.
  Interventions: Drug: nucleoside analog reverse transcriptase inhibitor

INTERVENTIONS:
Drug: nucleoside analog reverse transcriptase inhibitor — tablets 100mg qd
  Other Names: lamivudine

SUMMARY:
The aim of this study is to identify the incidence of hepatitis B virus reactivation rate in Diffuse Large B Cell or high grade Follicular lymphoma patients with prior resolved hepatitis B undergoing RCHOP immuno-chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Naive DLBCL or high grade FL patients
* Age range 18-75 years old
* ECOG performance status 0-3
* Life expectancy of more than 3 months
* Adequate organ function
* HBsAg negative/HBcAb positive at baseline

Exclusion Criteria:

* Infection of HAV,HCV,HIV
* Pregnant or lactating women
* Serious uncontrolled diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
incidence of HBV reactivation | from the first cycle of RCHOP (day 1) to six months after the last cycle of RCHOP
  HBV reactivation is defined as- the level of HBV-DNA exceeds the upper limit of normal(ULN).

SECONDARY OUTCOMES:
the outcome of antiviral therapy in HBV-DNA abnormal patients | from the initiation of antiviral thearpy to six months after the last cycle of RCHOP
  Once the level of HBV-DNA exceeds the upper limit of normal, antiviral therapy will be given immediately.Liver function and serum HBsAg and HBcAg of these patients will be monitored until six months after the last dosing of RCHOP.

CONTACTS AND LOCATIONS:
Overall Officials: Junning Cao, Doctor, Principal Investigator — member of Fudan University
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality